CLINICAL TRIAL: NCT06020846
Title: Comparison of the Immediate Effects of Soleus Pushup Exercise and Treadmill Walk on Blood Glucose Levels in Type 2 Diabetes Population.
Brief Title: Effect of Soleus Pushup Exercise in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Ume Farva
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus, type 2; soleus push up; treadmill walk; blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soleus Pushup Exercise group A (Experimental): soleus push up exercise
  Interventions: Other: Soleus Pushup Exercise
- Treadmill group 2 (Active Comparator): treadmill walk
  Interventions: Other: treadmill walk group 2

INTERVENTIONS:
Other: Soleus Pushup Exercise — Patient will be seated on a chair, his legs at 90 degrees to the floor, keep the toes, and feet flat on the ground, and move his heels up and down continuously.
  4 sets of 15 minutes each,1hour total intervention time
  Arms: Soleus Pushup Exercise group A
Other: treadmill walk group 2 — The patient will do treadmill walk at normal walking speed, 4 sets of treadmill walk for 15 minutes each, 1hour total intervention time
  Arms: Treadmill group 2

SUMMARY:
The aim of this research is to compare the immediate effects of one hour Soleus Pushup Exercise and treadmill walk in Type 2 Diabetic population on blood glucose level. Randomized controlled trials done at Railway General Hospital and diabetic centers of Rawalpindi and Islamabad.. The sample size was 66. The subjects were divided in two groups, 33 subjects in Soleus Pushup Exercise group and 33 subjects in treadmill walk group. Study duration was of 6 months. Sampling technique applied was non probability convenience sampling technique. Only 40-60 years diabetic people with clinically diagnosed type 2 Diabetes for upto 10 years were included. Tools used in the study are Glucometer

DETAILED DESCRIPTION:
Diabetes is on the rise worldwide, with a global prevalence in adults in 2021 being 537 million adults (20-79 years) living with diabetes -one in ten. This number is predicted to rise to 643 million by 2030 and 783 million by 2045. Over 3 in 4 adults with diabetes live in low- and middle-income countries. Although physical activity (PA) is a key element in the prevention and management of type 2 diabetes. Structured interventions combining Physical Activity and modest weight loss have been shown to lower type 2 diabetes risk by up to 58% in high-risk populations. The increase in T2DM prevalence can only partly be attributed to the increasing prevalence of obesity and a sedentary lifestyle. The exercise recommendations for individuals with type 2 diabetes are similar as for the general population, suggesting a minimum of 150 min of moderate-vigorous-intensity aerobic exercise each week. However, the general population doesn't adhere to these guidelines.

The goal of treatment in type 2 diabetes is to achieve and maintain optimal BG, lipid, and blood pressure (BP) levels to prevent or delay chronic complications of diabetes. A fundamental principle in exercise physiology is that a small muscle mass working in isolation can achieve a higher local oxygen consumption (VO2/min per kg) than when recruiting a large muscle mass. The soleus (1% body mass) has a highly pennated architecture favoring greater amounts of muscular work during plantarflexion. It has an exceptionally high physiological cross-sectional area (3-8 times more than most of the 20 other limb muscles studied).

ELIGIBILITY:
Inclusion Criteria:

* • Both male and female individuals

  * Individuals with age between 40 to 60 years
  * Individuals with clinically diagnosed diabetes type 2 up to 10 years
  * individuals not engaged in a structured walking/exercise program
  * 2 hours post meal with glucose ranging upto 200.

Exclusion Criteria:

* • No recent or planned changes in diet, physical activity, or medications.

  * Participants diagnosed with pre-diabetes, gestational diabetes, or type 1 diabetes

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | baseline to 30 minutes and 60 minutes
  The blood glucise level will be measured by the glucometer at base line , 30 min and at 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No